CLINICAL TRIAL: NCT06756165
Title: Community-Based Mental Health Screening & Referral for Flood-Affected Women in Dadu: A Feasibility Study
Brief Title: Community Based Mental Health Screening and Referral
Acronym: MeSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Jai Kumar Das (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor-Investigator, Dr Jai Kumar Das, Associate Professor and Assistant Director, Aga Khan University
Organization: Aga Khan University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-10475-30776; 53600 (Other Grant/Funding Number: Grand Challenges Canada)
Record Dates: First submitted 2024-12-20; First posted 2025-01-01 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Mental Health; Depression; Anxiety Disorders; Community Health Services; Women's Health
Keywords: Mental Health Screening; Flood-Affected Women; Mental Health Referral; Mental Health Support; Screening and Referral Program; Health Services Accessibility
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study will adopt a parallel, quasi-experimental design with women of reproductive age in flood-affected areas of Dadu district. Participants will be purposively assigned to intervention or control groups. The intervention will include screening using PHQ-2 and GAD-2, followed by PHQ-9 and GAD-7 if positive, group awareness sessions, and referral to BHUs for care by trained psychologists or medical officers. Severe cases will be referred to tertiary care. Services will be delivered by trained LHWs, with one-time transport support. The control group will receive standard care without the mental health intervention. Both groups will be assessed at baseline and endline to compare changes in mental health status, service use, and care-seeking behavior.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): This arm focuses on enhancing mental health through structured activities integrated into existing community and primary health services. Participants in this arm will receive additional support to address mental health challenges within the flood-affected communities of Dadu. The intervention leverages trained Lady Health Workers (LHWs) and healthcare staff at primary health centers to screen, manage and provide timely referrals.
  Interventions: Behavioral: Mental health screening
- Control Arm (No Intervention): Participants in the control arm will receive the standard care currently provided in the study area, which includes routine health services delivered by community health workers and the healthcare system. The control arm serves as a comparison group, enabling an evaluation of the additional impact of the intervention on mental health outcomes, resilience, and community engagement.

INTERVENTIONS:
Behavioral: Mental health screening — Participants in the intervention arm will receive a mental health screening, referral, and counselling program by trained LHWs and BHU staff. LHWs will screen 120-170 WRA using PHQ-2 and GAD-2. Screen-positive WRA will be referred to BHUs, where trained doctors will reassess them using PHQ-9 and GAD-7. Those with mild to moderate anxiety or mild to moderately severe depression will receive two counselling sessions (initial and follow-up), each lasting at least 20 minutes, covering psychoeducation, awareness, and coping strategies. Severe cases will be referred to tertiary care for specialized mental health services. Mild cases will be advised to join resilience-building sessions. All WRA will attend two of three monthly group sessions by LHWs (20-25 WRA, 2 hours each), focusing on mental health literacy and coping strategies, including those related to climate change stressors like floods.
  Arms: Intervention Arm

SUMMARY:
This feasibility study aims to evaluate the implementation of a community-based mental health screening, referral, and resilience-building intervention for flood-affected women of reproductive age (WRA) in a rural district of Dadu, Sindh, Pakistan. The quasi-experimental study uses a comparison group and involves training Lady Health Workers (LHWs) to conduct mental health screening using GAD-2 and PHQ-2 tools, refer screen-positive women to Basic Health Units (BHUs) for further assessment, and conduct group sessions on mental health awareness and climate resilience. BHU doctors will reassess referred women using GAD-7 and PHQ-9, provide psycho-counseling, and refer severe cases to tertiary care. The study will assess feasibility, acceptability, appropriateness, and effectiveness of the intervention to inform scalable mental health strategies for disaster-prone settings.

DETAILED DESCRIPTION:
This study evaluates the feasibility and implementation of a community-based mental health screening, referral, and resilience-building intervention for women of reproductive age (WRA) affected by the 2022 floods in the Dadu district of Sindh, Pakistan. The intervention engages Lady Health Workers (LHWs) to screen WRA using validated tools-GAD-2 and PHQ-2. Women scoring ≥3 on either scale will be referred to Basic Health Units (BHUs), where trained facility-based doctors will reassess them using the GAD-7 and PHQ-9 instruments. Based on the diagnosis, WRA with mild to moderate symptoms will receive two structured counseling sessions, while those with severe symptoms will be referred to tertiary care with logistical support.

In parallel, LHWs will conduct monthly group sessions to raise mental health awareness, address stigma, and build community resilience to climate change-related hazards such as flooding. These sessions, based on a standardized curriculum, are open to all WRA regardless of screening status and focus on stress management, coping strategies, and emotional support.

The study employs a quasi-experimental design with a comparison group across selected union councils. The intervention will be evaluated through baseline and end-line quantitative surveys as well as qualitative assessments via focus group discussions (FGDs) and in-depth interviews (IDIs). The primary outcomes include feasibility, acceptability, appropriateness, and awareness levels, while the secondary outcome assesses the effectiveness of the intervention in reducing symptoms of depression and anxiety.

The findings will guide future efforts to integrate mental health services into primary care and community-based disaster preparedness strategies in Pakistan and similar contexts.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age (WRA) 18-49 years in the targeted area

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only individuals who self-identify as female are eligible to participate in this study.
Enrollment: 4800 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of Intervention | Data will be collected at baseline and approximately 12 months after the intervention begins.
  A structured questionnaire will be used to assess the feasibility of implementing the community-based mental health screening, referral, and resilience-building intervention. It will be administered to Lady Health Workers (LHWs), health facility staff, and program implementers. The tool will assess recruitment success, retention rates, adherence to protocol, and challenges encountered during implementation.
  Measurement Tool: A specifically designed feasibility assessment questionnaire.

SECONDARY OUTCOMES:
Anxiety Symptoms | Assessed at baseline and 12 months after intervention initiation.
  Anxiety symptoms will be measured using the Generalized Anxiety Disorder-7 (GAD-7), a validated screening tool. Scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms.
  Measurement Tool: GAD-7 questionnaire.
Depression Symptoms | Assessed at baseline and 12 months after intervention initiation..
  Depression symptoms will be assessed using the Patient Health Questionnaire-9 (PHQ-9), a standardized and validated tool. Scores range from 0 to 27, with higher scores reflecting greater severity.
  Measurement Tool: PHQ-9 questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sinddh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon individual reasonable requests, subject to approval from the institute and funders, and following the establishment of a formal data transfer agreement.

REFERENCES:
- [Derived] Das JK, Gaffey MF, Ansari ZN, Mirani M, Tabassum F, Niaz M, Siddiqui A, Rabbani F, Rizvi A, Ahmed I, Khan M, Bhutta ZA. Community-based mental health screening & referral for flood-affected women in rural Pakistan: an intervention feasibility study protocol. BMJ Open. 2025 Oct 23;15(10):e104759. doi: 10.1136/bmjopen-2025-104759. PMID 41130670